CLINICAL TRIAL: NCT01462409
Title: Luftfeuchtigkeit Unter CPAP Mit Temperatur- Und Feuchtigkeitskontrolle
Brief Title: Humidity Under Continuous Positive Airway Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: ResMed GmbH & Co KG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Climateline2011
Record Dates: First submitted 2011-10-20; First posted 2011-10-31 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Sleep Apnea, Obstructive
Keywords: obstructive sleep apnea; humidification; mask; heated tubing
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Humidifiers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- heated humidification (Experimental)
  Interventions: Device: CPAP with heated humidification
- No Humidification (Experimental)
  Interventions: Device: CPAP without humidification
- Controlled heated Humidification with heated tube (Experimental)
  Interventions: Device: RESMed S9 with humidifier H5i and heated tube Climate Line

INTERVENTIONS:
Device: RESMed S9 with humidifier H5i and heated tube Climate Line — At stable ambient room temperature and different CPAP pressure levels, 8 and 12 cmH2O, with and without additional leakage, humidity and temperature is measured inside of a patients nasal mask. Controlled heated humidification with heated tubing (Climate Line).
  Arms: Controlled heated Humidification with heated tube
Device: CPAP without humidification — At stable ambient room temperature and different CPAP pressure levels, 8 and 12 cmH2O, with and without additional leakage, humidity and temperature is measured inside of a patients nasal mask. Without any humidification.
  Other Names: ResMed S9 without humidifier
  Arms: No Humidification
Device: CPAP with heated humidification — At stable ambient room temperature and different CPAP pressure levels, 8 and 12 cmH2O, with and without additional leakage, humidity and temperature is measured inside of a patients nasal mask. With controlled heated humidification and standard tubing.
  Other Names: RESMed S9 with humidifier H5i
  Arms: heated humidification

SUMMARY:
Heated humidification in CPAP therapy is often not enough to prevent side effects like dryness of nasal mucosa and xerostomia, especially in cases of mouth breathing or mask leakage. Additionally a higher level of humidification in lower ambient room temperature can lead to condensation and irritating noises. Compliance of affected patients decreases considerably. Regarding this, devices with humidifier and additional heated tubing are developed to automatically regulate optimal humidification and temperature right up to the mask. The efficacy of a system with controlled heated humidification and heated tubing in nasal masks under various conditions like leakage and different pressure levels is object of this study.

DETAILED DESCRIPTION:
Participants will breath 3 hours during daytime with a nasal mask under three different humidity modes (No humidity, controlled heated humidification, controlled heated humidification with heated tubing) with CPAP 8 and 12 mmHg and with and without leakage. The ambient room temperature is controlled with air conditioning. Changes in temperature and humidity is measured inside of the mask with a humidity sensor and recorded. After each phase the participants subjective opinion about humidity and temperature is asked.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70
* Obstructive Sleep Apnoea Syndrome

Exclusion Criteria:

* Other severe acute or chronic nasal disease (rhinitis, sinusitis), Cardiovascular disease, respiratory or neurologic disease
* Incapable of giving consent

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Humidity differences | 3 hours per patient
  Changes of humidity and temperature under different conditions (e.g. with and without humidifier, leakage, pressure changes) measured breath by breath with humditiy sensor inside of a nasal mask.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Heinz Ruehle, MD, Principal Investigator — Institut für Pneumologie Hagen Ambrock eV
Locations (1):
- Helios Klinik Hagen Ambrock, Hagen, North Rhine-Westphalia, Germany